CLINICAL TRIAL: NCT02705547
Title: Open-label Biomarker Study of Rosuvastatin (Crestor) for the Treatment of Patients With Friedreich Ataxia
Brief Title: Rosuvastatin (Crestor) in Friedreich Ataxia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-012659
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Crestor) (Experimental): This is an open-label study of Rosuvastatin (Crestor) in patients with FRDA. Study subjects will receive 10 mg of Rosuvastatin daily for 3 months.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Daily oral administration of Rosuvastatin (10 mg) for 3 months
  Other Names: Crestor

SUMMARY:
This study is an exploratory open-label clinical trial of Rosuvastatin in patients with Friedreich ataxia (FRDA). This is an outpatient trial with the goal of enrolling 10 evaluable adults with genetically confirmed FRDA who are between the ages of 18-65. Subjects will receive 10mg of oral Rosuvastatin daily for three months.

DETAILED DESCRIPTION:
Friedreich ataxia (FRDA) is a progressive neurodegenerative disease of children and adults for which there is presently no therapy. Much of the current work in FRDA is aimed at finding new targets for drug therapies. Recent work at the University of Pennsylvania has discovered that serum ApoA-1 protein levels are lower in people with FRDA when compared with control levels. ApoA-1 is the main protein found in high-density lipoprotein (HDL) cholesterol and individuals with FRDA frequently have low HDL levels; the current study proposes to assess if administration of HMG-CoA reductase inhibitors for 3 months alters ApoA-1 protein levels in FRDA. Although the significance of ApoA-1 levels among FRDA patients is currently unknown, this study is proposed as an exploratory study to further examine this protein. If ApoA-1 protein levels increase over the course of treatment, future studies may additionally focus on examining this as a potential therapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Friedreich Ataxia confirmed by genetic testing
* Adults between the ages of 18 and 65
* Stable quinone dose (at least 1000 mg of Idebenone or 200 mg Coenzyme Q10) for 14 days prior to study entry and for the duration of the study
* Females who are not pregnant or breast feeding, and who do not intend to become pregnant.
* Subject has voluntarily signed consent form
* Willingness and ability to comply with all study procedures

Exclusion Criteria:

* Treatment with statins during the six previous months before study inclusion
* Currently active or unresolved liver or kidney disease
* Known history of renal insufficiency or creatine kinase >2 x ULN
* Use of red rice yeast during the previous six months before inclusion
* Current use of niacin and/or fibric acid derivatives
* Current use of cyclosporine
* Use of any investigational product within 30 days of baseline visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Change in ApoA-1 serum protein levels from baseline to Week 12 visit | 12 weeks
  Serum ApoA-1 protein levels will be collected at baseline and again at the Week 12 visit.

SECONDARY OUTCOMES:
Change in frataxin levels from baseline to Week 12 visit | 12 weeks
  Frataxin levels in whole blood and buccal cells will be collected at baseline and again at the Week 12 visit.
Change in platelet metabolism from baseline to Week 12 visit | 12 weeks
  Platelet metabolism will be assessed by performing liquid chromatography-mass spectrometry analysis on whole blood samples collected at baseline and again at the Week 12 visit.

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, MD PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No